CLINICAL TRIAL: NCT07018362
Title: Research on the Application of Ultrasonography in Fetal Growth Parameters
Brief Title: Ultrasound Assessment of Fetal Growth Parameters
Status: Enrolling by invitation | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, YiMing Su, Director, The First Affiliated Hospital of Xiamen University
Other Study IDs: FirstAHXiamenUsym
Record Dates: First submitted 2025-06-03; First posted 2025-06-12 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Fetal Clavicle Length; Fetal Scapular Width; Fetal Sternal Length; Fetal Scapular Length; Perinatal Outcomes of the Mother and Fetus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: restricted fetal growth — The fetus is of abnormal size and has not reached its genetic growth potential in utero. Fetal birth weight is less than two standard deviations from the average weight for the same gestational age, or less than the 10th percentile of normal weight for the same age.

SUMMARY:
The goal of this observational study is to establish reference value ranges for normal fetal biometric parameters at different gestational weeks for the domestic population, and evaluate their clinical application to predict perinatal outcomes. The main question it aims to answer is:

What is the relationship between fetal parameter measurements (such as clavicle length, scapular width, scapular length, sternum length, and cranial structure measurements) and gestational age as well as other growth parameters?

And how can these parameters be used in clinical applications such as predicting perinatal outcomes?

Researchers will observe the relationship between the measurement values of fetal clavicle length, scapular width, scapular length, sternum length, and cranial structure and gestational age as well as other growth parameters, and ultimately follow up on the perinatal outcomes of mother and fetus.

ELIGIBILITY:
Inclusion Criteria:

Singleton pregnancy; The date of the last menstrual period was determined for each pregnant woman, and a history of regular menstrual cycles was confirmed; Pregnant women had no maternal diseases that could affect fetal growth and development, such as diabetes, pregnancy-induced hypertension, or chronic infections; Fetuses had no chromosomal or structural abnormalities; Gestational age (calculated based on the last menstrual period) was within 7 days of the ultrasound biometric measurements; Good image quality.

Exclusion Criteria:

Multiple gestation, fetal demise, or stillbirth; Pregnancy complications or comorbidities affecting fetal growth; Clinically diagnosed fetal growth restriction (FGR); Confirmed pathogenic infections (serology-positive), including TORCH, HIV, RPR, or other infections; Prenatal ultrasound indicating fetal hydrops, structural anomalies, or chromosomal abnormalities; History of substance abuse (e.g., drugs, smoking, alcohol) or medication use in early pregnancy; Discrepancy between clinical gestational age and ultrasound-estimated gestational age; Lack of follow-up information.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women with singleton pregnancies at 12 to 40 weeks of gestation
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
fetal clavicle length | gestational weeks 12 to 40
  By sliding the probe at the fetal thoracic inlet, the clavicle can be visualized. Continuously adjust the probe orientation during scanning to ensure the clavicle is displayed at its maximum length. Place the electronic calipers at the midpoint of the sternal end and the acromial end of the clavicle, respectively. The measured distance represents the clavicular length, expressed in centimeters (cm).
scapular width and scapular length | gestational weeks 12 to 40
  Identify the fetal spine in the longitudinal plane. Align the probe parallel to this plane and move it laterally, continuously adjusting and slightly rotating the probe until the acoustic window simultaneously displays both the acromion and inferior angle of the scapula. The maximum distance between these two landmarks represents the scapular length.
  For scapular width measurement: Based on the scapular length view, further rotate the probe centered on the acromion to approximate a transverse fetal plane until the scapular spine is fully visualized at its maximal length. The longest distance between the acromion and medial border of the scapular spine is defined as the scapular width. All measurements are expressed in centimeters (cm).
sternal length | gestational weeks 12 to 40
  On the coronal or sagittal plane of the fetal chest region, continuously adjust the probe until the full length of the fetal sternum is visualized. Place the electronic calipers at the cephalic end of the first ossification center and the caudal end of the last ossification center, respectively. The measured distance represents the sternal length, expressed in centimeters (cm).

CONTACTS AND LOCATIONS:
Locations (1):
- EPIQ 7 (Philips Healthcare, Bothell, WA) 和 Voluson E10 (GE Healthcare, Milwaukee, WI), Xiamen, Fujian, China